CLINICAL TRIAL: NCT00788801
Title: Exploratory Positron Emission Tomography (PET) Study to Evaluate the Effects of ABT-614 on [11C]-(+)-PHNO Binding Potential to D3 Receptors in the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Beatrice Rendenbach-Mueller, PhD/Project Director, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M10-423
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-09

CONDITIONS: Healthy Volunteers

ARMS (3):
- Baseline (Experimental)
  Interventions: Drug: ABT-614
- ABT-614 Low Dose (Experimental)
  Interventions: Drug: ABT-614
- ABT-614 High Dose (Experimental)
  Interventions: Drug: ABT-614

INTERVENTIONS:
Drug: ABT-614 — Baseline PET scan with radiotracer only, PET scan with radiotracer and ABT-614 Low Dose or ABT-614 High Dose

SUMMARY:
This study is being done in healthy volunteers to help researchers understand how ABT-614 works in the human body, specifically in the brain. The PET imaging technique can be thought of as a way to take pictures of chemical changes in the brain. To take a PET scan (picture), a substance with low levels of radioactivity (radiotracer) has to be injected when you are in the PET camera. The radiotracer is only radioactive for a short period of time. In this study, PET is being used to measure how the study drug attaches to specific receptors in the brain. The radiotracer used in this study, [11C]-(+)-PHNO, is currently being used for studies in people at the CAMH PET Centre.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) is 18 to 26 kg/m2, inclusive
2. A condition of general good physical health based upon the results of a medical history, physical examination, vital signs, laboratory profile, 12-lead electrocardiogram (ECG)

Exclusion Criteria:

1. Presence of a metal implant (i.e., aneurysm clip, metal fragments, internal electrical devices such as a cochlear implant, spinal cord stimulator or pacemaker) that would preclude a MRI scan
2. During the last year, a radiation exposure that on its own or in addition to the expected radiation from this study exceeds the allowed annual radiation exposition level (20 mV)
3. Use of tobacco or other nicotine-containing products within 6 months prior to Screening
4. Diagnosis of substance or alcohol disorder within 12 months prior to Screening
5. History of claustrophobia or feeling of inability to lie still on his back in the PET camera
6. History or presence of any neurological or psychiatric conditions

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
D3 receptor occupancy as estimated by measuring ABT-614 induced changes in [11C]-(+)-PHNO BP | At the approximate Tmax following a single dose of study drug

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Site Reference ID/Investigator# 12201, Toronto, Ontario
  - Site Reference ID/Investigator# 13961, Toronto, Ontario